CLINICAL TRIAL: NCT07043088
Title: The SWEEP Trial - Serial Versus no Membrane Sweeping on Spontaneous Onset of Labor: a Randomized Controlled Trial
Brief Title: The SWEEP Trial: a Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-10-72-82-24
Record Dates: First submitted 2025-06-11; First posted 2025-06-29 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-06

CONDITIONS: Membrane Stripping; Cervical Ripening; Memrane Sweeping
Keywords: membrane sweeping; cervical ripening; labor onset; term pregnancy; induction of labor; midwifery; randomized controlled trial; post-term pregnancy; membrane stripping
MeSH Terms: conditions — Pregnancy, Prolonged

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No membrane sweeping (No Intervention): Participants allocated to the control group will receive standard antenatal care, which does not include membrane sweeping prior to gestational age 41+3.
- Membrane sweeping (Experimental): Participants allocated to the intervention group will receive standard anetnatal care plus serial membrane sweeping starting from the time of allocation at gestational age 39+5 to 40+2. A total of up to three membrane sweepings will be scheduled, each with an interval of 2-3 calendar days
  Interventions: Procedure: Membrane sweeping

INTERVENTIONS:
Procedure: Membrane sweeping — Serial membrane sweeping from gestational age 39+5-40+2 with 2-3 days interval and a maximum og three times.
  Other Names: Intervention group
  Arms: Membrane sweeping

SUMMARY:
The purpose of this clinical trial is to determine whether serial membrane sweeping at term is more effective than no membrane sweeping in promoting spontaneous onset of labor.

The primary research question is whether serial membrane sweeping increases the likelihood of birth before gestational age 41+3 with spontaneous onset of labor.

A total of 1536 participants will be randomized between gestational age 39+5 and 40+2 to either no membrane sweeping or up to three membrane sweepings performed 2-3 days apart.

Researchers will collect data from the electronic medical record and participants will be asked to complete a short daily questionnaire on pregnancy symptoms and, in the intervention group, their experience of membrane sweeping from randomization until birth. All participants will be asked to complete a follow-up questionnaire about their birth experience five weeks postpartum

DETAILED DESCRIPTION:
Background and Objective:

Membrane sweeping is a simple mechanical procedure used at term to promote spontaneous onset of labor by stimulating local prostaglandin release. Although it is widely used and generally considered safe, evidence for its effectiveness is limited and of low certainty. The SWEEP trial is a multicenter randomized controlled trial designed to address this gap by investigating whether serial membrane sweeping starting between GA 39+5 and 40+2 increases the likelihood of spontaneous labor before GA 41+3 compared to no membrane sweeping.

Study design:

This is a pragmatic, open-label, multicenter, randomized controlled trial conducted in public antenatal clinics in Denmark. A total of 1536 pregnant women with low-risk, singleton pregnancies will be randomized between GA 39+5 and 40+2 to either: No membrane sweeping, or serial membrane sweeping with 2-3 days interval, max. three times.

Intervention and Procedures:

If possible, the first membrane sweeping will be performed during the routine antenatal visit at term. If not feasible, a separate consultation will be arranged. Two additional appointments will be scheduled as needed. Membrane sweeping is performed by inserting one or two fingers through the cervix and rotating them 2-5 times to separate the fetal membranes from the lower uterine segment. If the cervix is closed, cervical massage is performed externally with circular motions for approximately 15 seconds.

The intervention will continue until spontaneous labor begins or a maximum of three sweepings have been performed.

Participants in the control group will receive routine midwifery care but will be asked to avoid membrane sweeping until at least GA 41+3, unless medically indicated.

Inclusion criteria:

Singleton pregnant women at term with a fetus in cephalic presentation and an intended vaginal delivery.

Exclusion criteria:

< 18 years of age Unable to speak and understand Danish Gestational age not determined by Crown-Rump-Length Previous cesarean section Ruptured membranes Painful contractions Vaginal bleeding more than bloody discharge Membrane sweeping performed within the last two weeks Already scheduled IOL or any known indication for IOL at or prior to GA 41+3 based on local or national guidelines Known low-lying placenta (placenta located <3 cm from the internal orifice verified by transvaginal ultrasound)

Outcomes:

The primary outcome is birth < GA 41+3 with spontaneous onset of labor.

Key secondary outcomes:

Risks and Side Effects:

There are no known serious risks associated with membrane sweeping for either the mother or baby.

Common and mild side effects may include:

Discomfort or mild pain during the procedure (the procedure can be stopped at any time upon request) Light spotting or brown discharge Braxton Hicks contractions

Informed Consent and Ethical Considerations:

Participants will receive both oral and written information in accordance with national and international ethical guidelines. Consent is obtained digitally via the REDCap platform using secure electronic signature technology.

Participants may withdraw consent at any time without consequence. All data are processed in accordance with the Danish Health Act and applicable GDPR regulations.

The study has been approved by the Regional Committees on Health Research Ethics for Central Denmark Region (journal number: 1-10-72-82-24 ) in accordance with Danish law and the Declaration of Helsinki.

Funding:

Funding for the trial is donated by:

Sundhedsdonationer from the Danish health insurance "danmark" with 7,000,000 DKK, The Health Research Foundation of Central Denmark Region with 100,000 DKK The Danish Association of Midwives with 45,931 DKK.

Additional funds will be sought to cover running costs during the trial. The investigators have no financial interests in the funding organizations.

Dissemination:

Study results will be published in international peer-reviewed journals and made publicly accessible in accordance with transparency requirements.

ELIGIBILITY:
Inclusion Criteria:

Singleton pregnant women at term with a fetus in cephalic presentation and an intended vaginal delivery.

Exclusion Criteria:

* < 18 years of age
* Unable to speak and understand Danish
* Uncertain gestational age , defined as gestational age not determined by Crown-Rump-Length
* Previous cesarean section
* Ruptured membranes
* Painful contractions
* Vaginal bleeding more than bloody discharge
* Membrane sweeping performed within the last two weeks
* Already scheduled IOL or any known indication for IOL at or prior to GA 41+3 based on local or national guidelines
* Known low-lying placenta (placenta located <3 cm from the internal orifice verified by transvaginal ultrasound)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1536 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Spontaneous Onset of Labor Resulting in Birth Before 41+3 Weeks of Gestation | From randomization until time of birth. Assessed at birth
  Participants meet the primary outcome if they give birth before gestational age 41 weeks and 3 days, and labor starts spontaneously-defined as either prelabor rupture of membranes (PROM) or contractions leading to cervical dilation, without the use of medical or mechanical induction methods (including artificial rupture of membranes before 4 cm dilation) and without a cesarean section before labor begins

SECONDARY OUTCOMES:
Undelivered at Gestational Age 41+3 | From randomization until time of birth. Assessed at birth.
  Still pregnant when entering the calendar date of GA 41+3 (deliveries at 41+3 counts as undelivered)
Gestational Age at Delivery | From randomization until time of birth. Assessed at birth
  Length of gestation at birth in days
Randomization to Delivery Interval | From date of randomization until the date of birth, assessed up to 21 days
  Hours from randomization to birth
Duration of Labor | From onset of labor (self-reported contractions or spontaneous rupture of membranes) until time of birth.
  Hours from selfreported starting time of contractions or spontaneous rupture of membranes till time of birth
Duration of Active Labor | From active phase of labor to time of birth
  Minutes from active phase of labor registered in the electronic medical journal to time of birth or minutes from 4-6 cm of cervical dilation and painful contractions to time of birth.
Induction Of Labor (IOL) | From date of randomization until time of birth. Assessed within 21 days.
  Labor started with any induction method including AROM <4 cm
Indication for Induction of Labor | From date of randomization until time of birth. Assessed within 21 days.
  IOL due to:
  * Late term pregnancy (from GA 41+3-)
  * Maternal request
  * Maternal medical indication
  * Fetal indication
  * Other indications
Spontaneous Rupture of Membranes | From date of randomization until time of birth. Assessed within 21 days.
  Spontaneous rupture of membranes as primary labor onset occurring before contractions
Use of Oxytocin Augmentation | From active phase of labor to time of birth
  Use of oxytocin augmentation during labor from more than 4 cm of cervical dilatation
Intrapartum Temperature equal to or greater than 38.0 degrees Celsius | From labor onset to time of birth
  Two rectal temperature measurements of 38.0 degrees Celsius or higher, taken at least 30 minutes apart
Epidural Analgesia During Labor | From labor onset to time of birth
  Administration of epidural from onset of labor till time of birth
Mode of Delivery | From onset of labor to time of birth
  Spontaneous vaginal delivery; no use of vacuum or forceps. Instrumental vaginal delivery: use of vacuum or forceps. Caesarean section: scheduled or acute
Early Labor Experience | 4-6 weeks postpartum
  Self-reported early labor experience measured using the validated Early Labor Experience Questionnaire (ELEQ); total and subscale scores calculated
Childbirth Experience | 4-6 weeks postpartum
  Self-reported childbirth experience measured using the validated Childbirth Experience Questionnaire (CEQ); total and subscale scores calculated.

OTHER OUTCOMES:
Method(s) used for Labor Induction | From date of randomization until time of birth. Assessed within 21 days.
  Method(s) used for labor induction:
  * Prostaglandin
  * oxytocin <4 cm of cervical dilatation
  * cervical ripening catheter
  * AROM
More than One Induction Method used | From date of randomization until time of birth. Assessed within 21 days.
  Use of >1 IOL method
Intrapartum Administration of Sntibiotics | From labor onset to time of birth
  Any antibiotics during labor
Endometritis Postpartum | From time of birth to 7 days postpartum
  Suspected or confirmed; requires hospital contact and antibiotics
Maternal Mortality | Randomization to 42 days postpartum
  Death of a female related to pregnancy or its management
Maternal Need for Intensive Care | Randomization to 7 days postpartum
  Admission to an ICU or a unit that provides 24-h medical supervision and is able to provide mechanical ventilation or continuous vasoactive drug support for pregnancy or childbirth related complications
Maternal Length of Hospital Stay | From time of birth to discharge from the hospital. Assessed within 42 days.
  Hours from admission to delivery ward to discharge
Postpartum hemorrhage | From labor onset until 2 hours postpartum.
  Total bleeding in ml. during delivery and up to 2 hours postpartum
Uterine Rupture | Randomization to time of birth
  Confirmed cases of uterine rupture
Abruptio Placentae | Randomization to time of birth
  Confirmed cases of abruptio placentae
Decreased Fetal Movements | Randomization to time of birth
  Hospital admission due to maternal concern over decreased fetal movements. Includes all cases leading to clinical assessment.
Telephone Consultations | Randomization to admission for delivery
  Telephone consultations defined as number of inquiries by telephone regarding a clinical pregnancy question from the woman to the delivery unit or antenatal clinic
Outpatient Visits | Randomization to admission for delivery
  Pregnancy-related outpatient visits not part of standard care or intervention
Hospital Admissions | Randomization to admission for delivery
  Pregnancy-related hospital admissions not part of standard care or intervention.
Perinatal Death | Randomization to 7 days postpartum
  Death within 7 days after birth, with specified type (antepartum, intrapartum, or neonatal), gestational age or age, and cause of death.
Serious Neonatal Morbidity | From time of birth until discharge from the hospital. Assessed within 42 days.
  Composite of serious neonatal morbidity including NICU admission, need for respiratory support, Apgar <7 at 5 minutes, acidemia, or sepsis.
Admission to Neonatal Intensive Care Unit | From time of birth until discharge from the hospital or within the first 72 hours postpartum
  Admission to NICU
Need for Respiratory Support | From time of birth until discharge from the hospital or within the first 72 hours postpartum.
  Need for respiratory support (intubation and mechanical ventilation, oxygen, continuous positive airway pressure (CPAP), or high-flow nasal cannula (HNFC)) within 72 hours after birth if admitted to a neonatal department.
Apgar score < 7 at 5 minutes | From time of birth until 5 minutes after birth. Assessed 5 minutes after birth.
  Apgar score < 7 at 5 minutes
Neonatal Acidemia | From time of birth to one hour postpartum
  pH < 7.10 in a sample of umbilical cord arterial blood or neonatal blood obtained within the first hour after birth.
Neonatal Sepsis | From time of birth until discharge from the hospital or within the first 72 hours postpartum
  Neonatal sepsis defined as antibiotic treatment continuously for 7 days minimum.
Membrane Sweeping Received Outside The Trial | From randomization until time of birth. Assessed 4-6 weeks postpartum
  Self-reported membrane sweeping performed outside the study protocol, e.g. by private provider or midwife via custom item in electronic questionnaire
Stated Preference for Future Membrane Sweeping | 4-6 weeks postpartum
  Self-reported stated preference for receiving membrane sweeping in a future pregnancy, reported via custom item in electronic questionnaire.
Term Pregnancy Symptoms | From date of randomization until date of birth. Assessed up to 15 days.
  Daily self-reported presence and severity of predefined term pregnancy symptoms using a custom electronic questionnaire.
Experience of Membrane Sweeping | From date of randomization until time of birth. Assessed up to three times within 7 days.
  Self-reported experience of membrane sweeping using a visual analogue scale (VAS) and supplementary custom items.
Number of membrane sweepings performed | From randomization until time of birth. Assessed up to 12 days.
  Total number of membrane sweepings performed
  * 0
  * 1
  * 2
  * ≥ 3
Number of cervical massages performed | Randomization to time of birth
  Total number of cervical massages performed
  * 0
  * 1
  * 2
  * ≥ 3

CONTACTS AND LOCATIONS:
Overall Officials: Julie Glavind, PhD, Associate Professor, MD, Principal Investigator — Aarhus University Hospital, Department of Obstetrics and Gynecology
Locations (1):
- Aarhus University Hospital, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data are available from the corresponding author upon reasonable request and in accordance with Danish data protection regulations.
Supporting Information: Study Protocol, SAP

REFERENCES:
- See also: The study's website — https://sweeptrial.dk/